CLINICAL TRIAL: NCT07036497
Title: THE IMPACT OF VITAMIN B12 TREATMENT ON EJACULATORY FUNCTIONS IN MEN: SYMPTOMATIC RELIEF AND IMPROVED OUTCOMES
Acronym: VITAMIN B12
Status: Completed | Type: Observational
Sponsor: OZGUR EKICI (Other)
Responsible Party: Sponsor-Investigator, OZGUR EKICI, MD, Erzincan Binali Yildirim Universitesi
Organization: Erzincan Binali Yildirim Universitesi (Other)
Other Study IDs: 2024-15/6
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Premature Ejaculation
Keywords: premature ejaculation, intravaginal ejaculatory latancy time, premature ejaculation diagnostic tool, vitamin B12, premature ejaculation profile
MeSH Terms: conditions — Premature Ejaculation | interventions — Vitamin B 12

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Vitamin B12 — Vitamin B12 treatment was initiated in male patients with vitamin B12 deficiency due to anemia etiology.

SUMMARY:
Aim: To investigate whether intramuscular B12 treatment has an effect on ejaculation in male patients with B12 deficiency.

Methods: Male patients who were diagnosed with vitamin B12 deficiency in the internal medicine outpatient clinic between October 2024 and March 2025 and started intramuscular B12 treatment were included in the study. The scores obtained from the self-estimated intravaginal ejaculation latency time (IELT), premature ejaculation diagnostic tool (PEDT) and premature ejaculation profile (PEP) questionnaires reflecting the ejaculatory status of these patients before treatment were recorded. After 3 months of treatment, these scores were re-recorded by phone call.

The scores recorded before and after treatment were compared. Results: The study included 54 patients. The mean age of the patients was 43.46±13.3 years, mean pretreatment IELT was 2.4±1.4 min, and mean pre-treatment PEDT score was 11.3±4.8. In both the whole patient group and the premature ejaculation (PE) group, a statistically significant difference was observed in the items of perceived control over ejaculation, satisfaction with sexual intercourse and interpersonal difficulty related to ejaculation from the PEP questionnaire form after treatment, no significant change was found in the item of personal distress related to ejaculation.

PEDT scores showed statistically significant improvement after treatment both in the whole patient group and in the PE group. In terms of IELT, no differences was observed in the whole patient group after treatment, whereas statistically significant improvement was observed in the PE group.

Conclusion: Intramuscular vitamin B12 may improve ejaculation times and satisfaction levels in patient's questionnaires forms in male patients.

ELIGIBILITY:
Male patients aged 18-70 years who were admitted to the internal medicine outpatient clinic between October 2024 and March 2025 with non-specific gastrointestinal complaints or to investigate the etiology of anemia and who were started on intramuscular vitamin B12 due to vitamin B12 deficiency were included in the study

-

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Male patients aged 18-70 years who were admitted to the internal medicine outpatient clinic of Bursa City Hospital between October 2024 and March 2025 with non-specific gastrointestinal complaints or to investigate the etiology of anemia and who were started on intramuscular vitamin B12 due to vitamin B12 deficiency were included in the study
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
intravaginal ejaculation latency time after treatment | 6 months
  intravaginal ejaculation latency time after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Nilufer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No